CLINICAL TRIAL: NCT06531512
Title: A Phase II/III Seamless Design, Randomized, Double-blind, Paralleled-group, Placebo-controlled Study to Evaluate the Efficacy and Safety of Xianglei Tangzu Gao for the Treatment of Wagner Grade II Diabetic Foot Ulcers
Brief Title: Evaluate the Efficacy and Safety of Xianglei Tangzu Gao for the Treatment of Wagner Grade II Diabetic Foot Ulcers
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oneness Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ON101CLCT06
Record Dates: First submitted 2024-07-26; First posted 2024-08-01 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Xianglei Tangzu Gao plus Standard of Care (Experimental): Xianglei Tangzu Gao will be applied twice daily for up to 16 weeks to the Target Ulcer.
  Interventions: Drug: Xianglei Tangzu Gao
- Vehicle Cream plus Standard of Care (Placebo Comparator): Vehicle cream will be applied twice daily for up to 16 weeks to the Target Ulcer
  Interventions: Other: Vehicle Cream

INTERVENTIONS:
Drug: Xianglei Tangzu Gao — Active ingredients: Extracts of Plectranthus amboinicus and Centella Asiatica
  Arms: Xianglei Tangzu Gao plus Standard of Care
Other: Vehicle Cream — Cream base of Xianglei Tangzu Gao
  Arms: Vehicle Cream plus Standard of Care

SUMMARY:
This is a phase II/III seamless design, randomized, double-blind, paralleled-group, placebo-controlled study to evaluate the efficacy and safety of Xianglei Tangzu Gao for the treatment of Wagner grade II diabetic foot ulcers. The primary endpoint is the proportion of subjects with complete closure of target ulcer during the 16-week treatment phase.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects, male or female, aged 18 to 80 years (inclusive) with Type 1 or Type 2 diabetes undergoing therapy for glycemic control using available diabetes drugs including insulin.
2. Subject has a glycosylated hemoglobin, HbA1c ≤ 12%.
3. Diagnosis with Diabetic Peripheral Neuropathy (DPN) or vascular disease defined by Chinese guidelines for diagnosis and treatment of diabetic foot (2020 version). Subject has adequate vascular perfusion of the affected limb, no obvious clinical manifestations of lower limb ischemia, confirmed by Ankle-Brachial Index (ABI) ≥ 0.8 and ≤ 1.3, or transcutaneous pressure of oxygen (TcPO2) > 30 mmHg on at least one lead.
4. An ulcer of Wagner Grade II.
5. Presence of at least one diabetic foot ulcer that meets all of the following criteria:

   1. Ulcer size (area) is > 1 cm2 and ≤ 25 cm2 (post-debridement at time of screening and randomization)
   2. Ulcer is located on or below the malleoli and presents duration of between 4 weeks and 12 months (at time of screening).
   3. If there are more than two ulcers, there should be a minimum 3 cm margin between the qualifying Target Ulcer and any other ulcers on the specified foot (post- debridement).
   4. No active infection by clinical inspection as defined by IDSA/IWGDF criteria. Note: If the subject has more than one qualifying diabetic foot ulcer, the most severe ulcer will be designated as the target ulcer. Severity will be determined by the investigator's assessment.
6. Subject, if a female of child-bearing potential, has a negative serum pregnancy test at screening, and willing to use 2 medically accepted methods of contraception (e.g., barrier contraceptives [female condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], and intrauterine devices) during the study (excluding women who are not of childbearing potential and/or who have been sterilized).
7. Subject should be able to walk and stand on the non-target ulcer limb.
8. Subject is willing to use an off-loading device for the target ulcer on the plantar while ambulation for the duration of the study
9. Subject and/or trained identified caregiver is able and willing to comply with study procedures and appropriate dressing changes.
10. A signed and dated informed consent form has been obtained from the subject prior to any study-related procedures being performed.

Exclusion Criteria:

1. In response to the standard of care, ulcer size reduction is > 30% during the two-week run-in Screening Period (between the first Screening Visit/V0 and Baseline/V2 randomization).
2. Ulcers with exposed bone or associated with osteomyelitis. Note: The osteomyelitis should be ruled out by clinical examination (probing of the wound) and X-ray findings.
3. Presence of necrosis, purulence, or sinus tracts that cannot be removed by debridement.
4. Laboratory values at Screening of:

   1. White Blood Cells (WBC) < 3.0 X 109 cells/L, > 12.0 X 109 cells/L
   2. C-Reactive Protein (CRP) >100 mg/L
   3. Liver function studies [Total bilirubin, aspartate aminotransferase (AST) and alanine transaminase (ALT)] > 3x the upper limit of normal
   4. Albumin < 25 g/L
   5. Renal function studies [Serum Creatinine] > 3x the upper limit of normal
   6. Hemoglobin< 100 g/L
5. Presence of any clinically significant medical condition(s) in medical history during screening period that, in the opinion of the investigator, could interfere with wound healing, including but not limited to the following:

   1. Acute or unstable Charcot foot
   2. Current sepsis
   3. Active malignant disease. A subject, who has had a malignant disease in the past, was treated, and is currently disease-free, may be considered for study entry.
   4. Acquired immune deficiency syndrome (AIDS) or HIV positive.
   5. Severe cerebrovascular lesion (acute or significant clinical manifestation) and severe cardiac dysfunction (NYHA class III or IV) such as congestive heart failure, myocardial infarction, or coronary artery bypass grafting, or percutaneous transluminal coronary angioplasty was performed within the last 6 months.
6. Subject is currently receiving (i.e., within 30 days of randomization visit) or scheduled to receive any of following medication or therapies, could interfere with wound healing during the study.

   1. immunosuppressants (including chronic systemic and topical steroids)
   2. cytotoxic chemotherapy
   3. cytostatic therapy
   4. negative pressure wound therapy
   5. autoimmune disease therapy
   6. dialysis
   7. lower limb revascularization surgery
   8. intravenous infusion of growth factors
   9. use of any investigational drug(s)
7. Previous use of bioengineered tissue or skin substitutes on potential target ulcers.
8. Subjects who need to stand continuously for more than 4 hours / day and have difficulty complying with off-loading instructions.
9. A psychiatric condition (e.g., suicidal ideation), current or chronic alcohol or drug abuse, determined from the subject's medical history, which, in the opinion of the investigator, may pose a threat to subject compliance.
10. Has any other factor which may, in the opinion of the investigator, compromise participation and/or follow-up in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with complete closure of Target Ulcer | 16-week Treatment Phase
  The primary efficacy endpoint for this study is the proportion of subjects with complete closure of Target Ulcer during the 16-week Treatment Phase, which is assessed by investigator.

SECONDARY OUTCOMES:
Time to complete closure of Target Ulcer | 16-week Treatment Phase
  Time to complete closure of Target Ulcer during the 16-week Treatment Phase, which is assessed by investigator.
The mean change for EQ-5D-5L score | Day 57, 85, 113 and 197
  The mean change for EQ-5D-5L score between baseline to Day 57, 85, 113 and 197
The proportion of subjects with complete closure of Target Ulcer | 16-week Treatment Phase
  The proportion of subjects with complete closure of Target Ulcer during the 16-week Treatment Phase, which is assessed by blinded independent review committee.

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ning, Principal Investigator — Ruijin Hospital
Locations (15):
- China (15):
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Shenyang Seventh People's Hospital (Shenyang Hospital of Integrated Traditional Chinese and Western Medicine), Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Nanfang Hospital, Guangzhou
  - Southern Medical University Third Hospital, Guangzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - Huadong Hospital Affiliated to Fudan University, Shanghai
  - Longhua Hospital Shanghai University of Traditional Chinese Medicine, Shanghai
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai TCM Integrated Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No